CLINICAL TRIAL: NCT04117178
Title: Monitoring Anti-Dementia Drugs by Serum Levels: Importance of Serum Levels, Drug-monitoring, Side-effects, Clinical Efficacy and Compliance (Translation of Official Danish Title)
Brief Title: Monitoring Anti-Dementia Drugs by Serum Levels
Acronym: MONANTI
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Zealand University Hospital (Other)
Collaborators: Filadelfia Epilepsy Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: REG-007-2018; 2017-002707-10 (EudraCT Number)
Record Dates: First submitted 2019-09-30; First posted 2019-10-07 (Actual); Results first posted 2025-02-10 (Actual); Last update posted 2025-02-10 (Actual); Status verified 2023-07

CONDITIONS: Dementia; Dementia With Lewy Bodies; Dementia in Parkinsons Disease; Dementia Alzheimers; Alzheimer Disease
Keywords: Therapeutic Drug Monitoring; TDM; Adverse effects; Dementia; Alzheimer's disease
MeSH Terms: conditions — Dementia; Lewy Body Disease; Alzheimer Disease | interventions — Donepezil; Memantine

STUDY DESIGN:
Intervention Model Description: Single blinded, randomized study with two arms: 'standard of care' arm and 'intervention' arm. Participants in the intervention arm will have their treatment adjusted according to Serum levels of the anti-dementia drug prescribed.
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard of care (Active Comparator): Participants allocated to this arm follow the usual routines of the out patient dementia clinic but are requested to have the serum level of the prescribed drug measured after 12 month. Also, CYP2D6, BcHE K and APOe4 status will be determined after 12 months.
  Interventions: Diagnostic Test: Measurement of serum level of anti-dementia drug
- Intervention arm (Experimental): Participants allocated to this arm follow are requested to inform the sponsor of any side effects up to 2 months after prescription of the anti-dementia drug. If so, they will have their treatment adjusted according to the serum level. Participants in the intervention arm not experiencing side effects will have their treatment adjusted after 6 months based upon serum level of the drug in question.
  Interventions: Drug: Donepezil; Drug: Memantine; Diagnostic Test: Measurement of serum level of anti-dementia drug

INTERVENTIONS:
Drug: Donepezil — Adjustment of treatment with donepezil according to serum level.
  Arms: Intervention arm
Drug: Memantine — Adjustment of treatment with memantine according to serum level.
  Arms: Intervention arm
Diagnostic Test: Measurement of serum level of anti-dementia drug — Participants allocated to the intervention arm are requested to inform the sponsor of any side effects up to 2 months after prescription of the anti-dementia drug. If so, they will have their treatment adjusted according to the serum level. Participants in the intervention group not experiencing side effects will have their treatment adjusted after 6 months based upon serum levels of the drug in question.
  Participants allocated to the standard of care arm follow the usual routines of the dementia clinic but are requested to have the serum level of the prescribed drug and CYP2D6-genotype measured after 12 month.

SUMMARY:
The main objective of the MONANTI study is twofold:

Firstly, to determine the serum concentration (SC) the anti-dementia drugs donepezil and memantine in a broadly defined clinical population of patients suffering from dementia treated with the two drugs in question. Secondly, to determine whether adjustment of treatment of anti-dementia medication based on measurements of the SC will benefit patients in terms of cognitive performance, activities of daily living (ADL), frequency and severity of side effects.

The reason for conduction of this study is that the relationship between serum-level of anti-dementia drugs, clinical efficacy, compliance and side effects has only been scarcely investigated.

Both a previously published study and a preliminary (pilot)study conducted imply that roughly 50 % of patients on donepezil have SC outside the recommended therapeutic reference range (TRR).

Thus, MONANTI will investigate if this is indeed the case in a broadly comprised population of patients with dementia treated with donepezil or memantine. In addition, MONANTI will link SC to co-morbidity, level of compliance, medication interactions. It is hypothesized that the efficacy of anti-dementia drugs can be significantly improved by adjustment of treatment according to SC. Also, it is hypothesized that the burden of side effects can be reduced in patients in whom too high SC are detected, if dose reduction or change of treatment drug is done.

MONANTI is a randomized study, in which the assessor is blinded to avoid related biases to the extent possible.

To meet the enrollment criteria eligible participants must:

A) be newly diagnosed with either Alzheimer's disease dementia, dementia with Lewy-bodies or Parkinson's disease with dementia and B) be scheduled for treatment with either donepezil or memantine. C) not meet a list of (exclusion) criteria, which have been set up in order to avoid blur and biases of the results.

D) be able to give written informed consent to participation in presence of a close relative.

After enrollment the participants will be randomly assigned to one of two study groups. In the first of these, the control group, the participants receive standard treatment and follow-up at the outpatient clinic. In addition, all participants in the control group who complete the trial will have a blood sample collected at the final visit to measure the SC of the anti-dementia drug along with a genetic test for a few key genes thought to be relevant for the study (two liver enzymes (cyp2D6, cyp3A4/5, APOE-genotype, butyrylcholine-esterase K-variant).

In the other group, the intervention group, the participators will be closely monitored for side effects after prescription of anti-dementia drugs. All participants in the intervention group will be offered a measurement of the SC in case they experience drug side effects within 2 months of treatment initiation. All participants in the intervention group will have a measurement of the SC done at the 6 months visit. The measured SC will be compared to the TRR of the drug in question. This information, along with details from the clinical assessment at the 6 month visit will be used to guide the decision of whether or not to adjust treatment. All decisions on treatment adjustment during the trial are done by the PI according to details in the protocol.

All participants in the intervention group are evaluated again at a 12 month visit, identical to that of the control groups.

To assess the possible effects of SC guided treatment adjustment six clinical tests/rating scales will be used (MMSE, ACE, NPI-Q, DAD, CGI, GDS). The tests/rating scales will be administered both at the enrollement visit and one year later at the final 12 month follow-up visit.

To measure the effect of donepezil on brain cholinergic function approx. 30 participants will be recruited for electroencephalography (EEG). These participants will have an EEG done at enrollment and after 12 months.

In addition to the above mentioned quantitative study a qualitative study with relatives of enrolled participants is planned.

All the needed approvals have been obtained according to Danish law (approval by the Danish Data Protection Agency, Scientific Ethics Committee for Region Sjaelland, The Danish Medical Agencies).

ELIGIBILITY:
Inclusion Criteria:

The following 3 inclusion criteria (A+B+C) must be met:

A. Participant must be newly diagnosed with one of the three conditions below

* Alzheimer's disease dementia
* dementia with Lewy Bodies
* Dementia in Parkinson's disease B. Participant must be prescribed either donepezil or memantine at enrollment. C. Participant must be able to give informed consent to participation in the study.

Exclusion Criteria:

* no accompanying relative at the enrollment and/or follow-up visits
* patients living alone who do not receive help to administer medication.
* lack of ability to cooperate, including severely reduced vision or impaired hearing and/or other severe disabilities.
* patients unable to give informed consent in a meaningful sense due to cognitive decline at enrollment.
* known psychiatric disease (schizophrenia, bipolar affective disorder etc.). However, patients suffering from depression are eligible if they have been in continuously medically treated for at least 3 months prior to enrollment.
* known neurologic disorder, which by it self could contribute to cognitive symptoms.
* other known medical condition (kidney-, liver-, metabolic disease etc.) which by itself could contribute to cognitive symptoms.
* treatment with anti-psychotic drugs within 3 months of possible enrollment. A minimal daily dosage of benzodiazepine is deemed permissable for enrollment.
* patients with a history of substantial previous abuse of alcohol or drugs. Also, any kind of substance abuse within last 3 months.
* any previous severe trauma to the head or neuroinfections which could contribute to cognitive symptoms.
* electro convulsive treatment within last 3 months.
* anesthesia within last 3 months

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 132 (Actual)
Dates: Start 2020-02-04 (Actual); Primary Completion 2023-02-16 (Actual); Study Completion 2023-02-16 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Peter Høgh, MD, ph.d., Principal Investigator — Regionalt Videnscenter for Demens; Michael Fischer, MD, Study Director — Regionalt Videnscenter for Demens
Locations (1):
- Regionalt Videnscenter for Demens, Roskilde, Region Sjælland, Denmark

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Fischer MHF, Zibrandtsen IC, Johannsen P, Siersma V, Rasmussen JB, Larsen JB, Hogh P. Therapeutic drug monitoring for dose optimization in Alzheimer's disease and in dementia with Lewy bodies: A randomized single-blinded clinical trial. J Alzheimers Dis Rep. 2024 Nov 24;8(1):1516-1528. doi: 10.1177/25424823241289373. eCollection 2024. PMID 40034344

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 132 participants recruited because a total of 110 participants assessable at the 6 month visit were needed.
Groups:
- Standard of Care: Participants allocated to this arm follow the usual routines of the out patient dementia clinic but are requested to have the serum level of the prescribed drug measured after 12 month. Also, CYP2D6, BcHE K and APOe4 status will be determined after 12 months.
  Measurement of serum level of anti-dementia drug: Participants allocated to the intervention arm are requested to inform the sponsor of any side effects up to 2 months after prescription of the anti-dementia drug. If so, they will have their treatment adjusted according to the serum level. Participants in the intervention group not experiencing side effects will have their treatment adjusted after 6 months based upon serum levels of the drug in question.
  Participants allocated to the standard of care arm follow the usual routines of the dementia clinic but are requested to have the serum level of the prescribed drug and CYP2D6-genotype measured after 12 month.
- Intervention Arm: Participants allocated to this arm follow are requested to inform the sponsor of any side effects up to 2 months after prescription of the anti-dementia drug. If so, they will have their treatment adjusted according to the serum level. Participants in the intervention arm not experiencing side effects will have their treatment adjusted after 6 months based upon serum level of the drug in question.
  Donepezil: Adjustment of treatment with donepezil according to serum level.
  Memantine: Adjustment of treatment with memantine according to serum level.
  Measurement of serum level of anti-dementia drug: Participants allocated to the intervention arm are requested to inform the sponsor of any side effects up to 2 months after prescription of the anti-dementia drug. If so, they will have their treatment adjusted according to the serum level. Participants in the intervention group not experiencing side effects will have their treatment adjusted after 6 months based upon serum levels of the drug in question.
  Participants allocated to the standard of care arm follow the usual routines of the dementia clinic but are requested to have the serum level of the prescribed drug and CYP2D6-genotype measured after 12 month.
Period: Overall Study
Arm/Group | Standard of Care | Intervention Arm
Started | 65 | 67
Completed | 49 | 58
Not Completed | 16 | 9

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Standard of Care | Intervention Arm | Total
Number analyzed (Participants) | 65 | 67 | 132
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 7 | 9 | 16
  >=65 years | 58 | 58 | 116
Age, Continuous [Mean (Standard Deviation); unit: years] | 76.0 (8.0) | 74.4 (8.1) | 75.2 (8.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 37 | 21 | 58
  Male | 28 | 46 | 74
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 65 | 67 | 132
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  Denmark | 65 | 67 | 132

OUTCOME MEASURES:

1. Primary Outcome: Change of Mini Mental State Examination (MMSE) Test Result
Description: Widely used clinical test for brief assesment of cognitive function. Total score ranging from 0 (worst) to 30 (best).
Time Frame: 1 year (enrollment in study and at 1-year follow-up)
Measure: Mean (Standard Deviation); unit: difference in MMSE units on a scale
Arm/Group | Standard of Care | Intervention Arm
Number analyzed (Participants) | 49 | 58
difference in MMSE units on a scale | -0.27 (3.19) | -0.90 (3.56)

2. Primary Outcome: Change of Adenbrooke's Cognitive Examination (ACE) Test Result
Description: Widely used clinical test for assesment of cognitive function. The total score ranges from 0 (worst) 100 (best) and includes the score of the MMSE test (0-30).
Time Frame: 1 year (enrollment in study and at 1-year follow-up)
Measure: Mean (Standard Deviation); unit: difference in ACE units on a scale
Arm/Group | Standard of Care | Intervention Arm
Number analyzed (Participants) | 49 | 58
difference in ACE units on a scale | -3.76 (6.56) | -4.02 (9.01)

3. Primary Outcome: Percentage of Participants With a Serum Concentration Within the Therapeutic Reference Range (TRR) at 12 Month Follow-up Visit.
Description: Percentage of participans in each group with serum concentrations of the study drugs within the therapeutic reference range (TRR) at the 12 month follow-up visit.
  According to the 2017 AGNP consensus guidelines the TRRs are "ranges of drug concentrations in blood that specify a lower limit below which a drug induced therapeutic response is relatively unlikely to occur and an upper limit above which tolerability decreases or above which it is relatively unlikely that therapeutic improvement may be still enhanced" (Pharmacopsychiatry . 2018 Jan;51(1-02):9-62. doi: 10.1055/s-0043-116492. Epub 2017 Sep 14).
  Donepezil has a serum TRR of 50-75 nanograms per milliliter (ng/mL) and memantine has a serum TRR of 90-150 ng/mL.
Time Frame: Counted at the 12 month visit
Measure: Count of Participants; unit: Participants
Arm/Group | Standard of Care | Intervention Arm
Number analyzed (Participants) | 49 | 58
Participants
  Within TRR | 23 | 23
  Outside TRR | 26 | 35

4. Primary Outcome: Level of Compliance to Treatment
Description: The level to which the medication has been ingested as prescribed. Both the participant him/her self is questioned as is the primary relative. The level of compliance is rated as belonging to one of the four categories: 1) 'completely regular drug intake' (no missed daily doses within 6 months), 2 'regular drug intake' (less than 10 missed daily doses within 6 months), 3) 'less regular drug intake' (10 - 30 missed daily doses with 6 months), 4) 'irregular drug intake' (more than 30 missed daily doses within 6 months)
Time Frame: Level of compliance will be scored at the one year follow-up by both questioning the participant and the primary relative.
Measure: Count of Participants; unit: Participants
Arm/Group | Standard of Care | Intervention Arm
Number analyzed (Participants) | 49 | 58
Participants
  Completely regular | 48 | 55
  Regular | 1 | 1
  Less regular | 0 | 2
  Irregular | 0 | 0

5. Secondary Outcome: Change of Clinical Global Impression (CGI) Score Result
Description: The overall clinical impression of the clinical response to treatment as assessed by the investigator. Ranges from 1 (very much improved) to 7 (very much worse).
Time Frame: 1 year (enrollment in study and at 1-year follow-up)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Standard of Care | Intervention Arm
Number analyzed (Participants) | 49 | 58
score on a scale | 4.68 (1.06) | 4.62 (0.95)

6. Secondary Outcome: Change in Geriatric Depression Scale (GDS) Symptoms Score
Description: The Geriatric Depression Scale (GDS) is a questionaire administered by the investigator to the participant. GDS is used to assess symptoms of depression in the elderly. A 15 item version of the GDS is used with a score from 0 (best) to 15 (worst).
Time Frame: The GDS is administered to all participants at the both the baseline and 12-month follow-up visit.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Standard of Care | Intervention Arm
Number analyzed (Participants) | 49 | 58
units on a scale | -0.57 (2.47) | 0.79 (2.55)

7. Secondary Outcome: Change of Disability Assessment for Dementia (DAD) Score Result
Description: A questionaire filled in by the primary relative of the participant. DAD measures the impact of dementia symptoms on activities of daily living (ADL), including eating, dressing, personal hygiene. Total score ranges from 0 (worst) to 40 (best)
Time Frame: 1 year (enrollment in study and at 1-year follow-up)
Measure: Mean (Standard Deviation); unit: difference in DAD units on a scale
Arm/Group | Standard of Care | Intervention Arm
Number analyzed (Participants) | 49 | 58
difference in DAD units on a scale | -0.07 (0.13) | -0.10 (0.16)

8. Secondary Outcome: Change of Neuropsychiatric Inventory Questionnaire (NPI-Q) Score Result
Description: A questionaire filled in by the primary relative of the participant. NPI-Q measures the severity of neuropsychiatric symptoms of demented patients. The total score ranges between 0 (best) and (36 worst).
Time Frame: 1 year (enrollment in study and at 1-year follow-up)
Measure: Mean (Standard Deviation); unit: difference in NPI units on a scale
Arm/Group | Standard of Care | Intervention Arm
Number analyzed (Participants) | 49 | 58
difference in NPI units on a scale | 2.40 (6.34) | 1.30 (3.18)

9. Secondary Outcome: C2D6 Phenotype
Description: Cyp2D6 is the gene which expresses the enzyme CYP2D6. Donepezil is metabolized by CYP2D6.
Time Frame: For participants in the standard of care arm CYP2D6 status will be determined 1 year after enrollment. For participants in the intervention arm Cyp2D6 will be tested within 2 months if side effects are experienced, if not then after 6 months.
Measure: Count of Participants; unit: Participants
Arm/Group | Standard of Care | Intervention Arm
Number analyzed (Participants) | 49 | 58
Participants
  Ultrafast metabolizer | 0 | 1
  Extensive metabolizer | 42 | 49
  Intermediate metabolizer | 5 | 5
  Poor metabolizer | 2 | 3

10. Secondary Outcome: Genetic Test for BcHE K Variant
Description: BcHE butyryl cholinesterase (BChE), K variant.
Time Frame: For participants in the standard of care arm BcHE K variant status will be tested 1 year after enrollment. For participants in the intervention arm BcHE K variant status will be determined at the 6 month follow-up.
Measure: Count of Participants; unit: Participants
Arm/Group | Standard of Care | Intervention Arm
Number analyzed (Participants) | 49 | 58
Participants
  Wildtype/Wildtype | 29 | 37
  Wildtype/mutant | 18 | 18
  mutant/mutant | 2 | 3

11. Other Pre Specified Outcome: Genetic Test for APOe4 Allele Status.
Description: The APOe4 allele is linked to an increased risk of developing Alzheimer's disease.
Time Frame: For participants who complete the trial APOe4 allele status is assessed at the 1 year visit.
Measure: Count of Participants; unit: Participants
Arm/Group | Standard of Care | Intervention Arm
Number analyzed (Participants) | 49 | 58
Participants
  APOE2/APOE2 | 0 | 1
  APOE2/APOE3 | 1 | 1
  APOE2/APOE4 | 1 | 1
  APOE3/APOE3 | 10 | 17
  APOE3/APOE4 | 31 | 28
  APOE4/APOE4 | 6 | 10

ADVERSE EVENTS:
Time Frame: Adverse event data were collected for each participant from the date of enrollment until the day of completion, ie. approximately 1 year.
Description: Details on all adverse events were collected and recorded according to the ICH E6 (R2) GCP guidelines. The primary investigator assessed whether an adverse event was classified as serious (Serious Adverse Event, SAE) or non-serious (non-serious adverse event, AE) and whether the event was related to the study drugs or not. Details on non-related SAEs and AEs were con not collected and reported according to prespecified criteria, instead a detailed description was given in the case report file.
Arm/Group | Standard of Care | Intervention Arm
All-Cause Mortality (participants affected / at risk) | 2/65 | 2/67
Serious Adverse Events (participants affected / at risk) | 6/65 | 7/67
Other Adverse Events (participants affected / at risk) | 42/65 | 46/67
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Standard of Care (N=65) | Intervention Arm (N=67)
Cholecystitis (Hepatobiliary disorders) | 0 (0) | 1 (1)
Psychosis (Psychiatric disorders) | 1 (1) | 0 (0) — Capgra syndrome
Psychosis (Psychiatric disorders) | 0 (0) | 1 (1)
Death (Surgical and medical procedures) | 1 (1) | 0 (0) — Fall causing hip fracture, resulting in death
Death (Vascular disorders) | 0 (0) | 1 (1) — Cardiac failure, anaemia
Donepezil overdose (General disorders) | 1 (1) | 0 (0) — Donepezil overdose (20 mg. daily for approx. 2 weeks) due to mistanke on part of the participant/relative.
COVID-19 (Infections and infestations) | 0 (0) | 1 (1) — COVID-19 respiratory infection
COVID-19 (Infections and infestations) | 0 (0) | 1 (1) — COVID-19 infection
Hospitalization due to headache (Nervous system disorders) | 1 (1) | 0 (0) — Tension-type headache
synkope (Vascular disorders) | 0 (0) | 1 (1) — Orthstatic Syncope
Stroke (Nervous system disorders) | 0 (0) | 1 (1) — Hospitalized due to stroke. Later death due to stroke complications.
Death due to lung cancer with metastases (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) — Diagnosed with lung cancer with cerebral metasteses after enrollment in study
Antebrachium facture (Surgical and medical procedures) | 1 (1) | 0 (0) — Antebrachium facture due to fall (bike accident)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Standard of Care (N=65) | Intervention Arm (N=67)
various minor non-related events (General disorders) | 42 (42) | 46 (46) — various minor non-related events not meeting the criteria for SAE.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2022-04-19): https://cdn.clinicaltrials.gov/large-docs/78/NCT04117178/Prot_SAP_000.pdf
  • Informed Consent Form (2019-03-12): https://cdn.clinicaltrials.gov/large-docs/78/NCT04117178/ICF_002.pdf